CLINICAL TRIAL: NCT00579995
Title: A Prospective, Randomized Trial Comparing Oral N-Acetylcysteine and Intravenous Sodium Bicarbonate for the Prevention of Contrast-Induced Nephropathy in High-Risk Patients Undergoing Cardiac Catheterization
Brief Title: A Prospective, Randomized TrialComparing Oral N-Acetylcysteine and Intravenous Sodium Bicarbonate
Acronym: PROTECt
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Technical measurement problems led to unreliable or uninterpretable data.
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 0120-05-FB
Record Dates: First submitted 2007-12-18; First posted 2007-12-24 (Estimated); Results first posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-08

CONDITIONS: Nephropathy
Keywords: contrast induced nephropathy
MeSH Terms: conditions — Kidney Diseases | interventions — Acetylcysteine; Sodium Bicarbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- N-Acetylcysteine (Active Comparator): Oral N-Acetylcysteine 600 mg
  Interventions: Drug: Oral N-Acetylcysteine
- Sodium Bicarbonate (Active Comparator): Sodium bicarbonate 3 milliliter per kilogram per hour (3 mL/kg/hr) infused at 1 mL/kg/hr for 6 hours post-procedure
  Interventions: Drug: Sodium Bicarbonate

INTERVENTIONS:
Drug: Oral N-Acetylcysteine — 600 milligrams (mg)
  Other Names: N-Acetyl-L-Cysteine
  Arms: N-Acetylcysteine
Drug: Sodium Bicarbonate — 3 milliliters per kilogram per hour (mL/kg/hr) for one hour pre-procedure and infused at 1mL/kg/hr for 6 hours post-procedure
  Other Names: Sodium hydrogen carbonate; sodium acid carbonate; baking soda
  Arms: Sodium Bicarbonate

SUMMARY:
The purpose of this study is to compare the efficacy of oral N-acetylcysteine and intravenous sodium bicarbonate for the prevention of Contrast-Induced Nephropathy (CIN) after cardiac catheterization.

DETAILED DESCRIPTION:
It is thought that N-acetylcysteine may reduce the ability of generated oxygen free radicals to damage cells by scavenging them. N-acetylcysteine may also increase the biologic effects of nitric oxide by combining with nitric oxide to form S-nitrosothiol, a more stable form and potent vasodilator. It also increases the expression of nitric oxide synthesis and may improve blood flow. Oxidants activate a signal-transduction cascade and molecular response that may initiate the cell-death pathway. These pathways seem to be sensitive to the redox state of the cell and are inhibited by N-acetylcysteine, which promotes pathways that lead to repair and survival whenever cells are under oxidant stress.

ELIGIBILITY:
Inclusion Criteria: 19 years of age

* Baseline serum creatinine or
* Calculated creatinine
* Stable Renal Function
* Left Ventricular ejection fraction
* Non-pregnant, non-lactating females (all women of childbearing potential must have a negative serum pregnancy test. No contraception will be required
* Able to sign informed consent

Exclusion Criteria:

* Acute renal failure
* History of Kidney transplant
* Currently receiving N-acetylcysteine

  _ Contraindication of hypersensitivity to N-acetylcysteine or sodium bicarbonate
* Left ventricular ejection fraction
* Pregnant, lactating females
* Allergy to contrast dye

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2005-05-01 (Actual); Primary Completion 2010-04-08 (Actual); Study Completion 2010-04-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Shurmur, MD, Principal Investigator — University of Nebraska
Locations (1):
- Unversity of Nebraska Medical Center, Omaha, Nebraska, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 1, N-Acetylcysteine: Oral N-Acetylcysteine - 600 milligram (mg)
- 2, Sodium Bicarbonate: Sodium bicarbonate, 3 milliliters per kilogram per hour (3 mL/kg/hr) for one hour pre-procedure and infused at 1 mL/kg/hr for 6 hrs post-procedure
Period: Overall Study
Arm/Group | 1, N-Acetylcysteine | 2, Sodium Bicarbonate
Started | 18 | 23
Completed | 18 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 1, N-Acetylcysteine: Oral N-acetylcysteine - 600 mg
- 2, Sodium Bicarbonate: Sodium bicarbonate 3 mL/kg/hr for one hour pre-procedure and infused at 1 mL/kg/hr for 6 hours post-procedure.
- Total: Total of all reporting groups
Arm/Group | 1, N-Acetylcysteine | 2, Sodium Bicarbonate | Total
Number analyzed (Participants) | 18 | 23 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 15 | 25
  >=65 years | 8 | 8 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (3.8) | 60 (4.4) | 61 (4.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 12 | 18 | 30
Region of Enrollment [Number; unit: participants]
  United States | 18 | 23 | 41

OUTCOME MEASURES:

1. Primary Outcome: Compare the Effectiveness of Two Medications for Prevention of Contrast-induced Nephropathy
Description: Compare oral N-Acetylcysteine and intravenous sodium bicarbonate for the prevention of contrast-induced nephropathy in high-risk patients undergoing cardiac catheterization.
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: milligrams per deciliter
Groups:
- 1, N-Acetylcysteine: N-Acetylcysteine - 600 milligram (mg)
- 2, Sodium Bicarbonate: 3 milliliter per kilogram per hour (mL/kg/hr) for one hour pre-procedure and infused at 1mL/kg/hr for 6 hours post procedure
Arm/Group | 1, N-Acetylcysteine | 2, Sodium Bicarbonate
Number analyzed (Participants) | 18 | 23
milligrams per deciliter | NA (NA) — Technical problems with measurement leading to unreliable or uninterpretable data. | NA (NA) — Technical problems with measurement leading to unreliable or uninterpretable data.

ADVERSE EVENTS:
Time Frame: 5 years
Groups:
- 1, N-Acetylcysteine: Oral N-acetylcysteine 600 mg
- 2, Sodium Bicarbonate: 3mL/kg/hr for one hour pre-procedure and infused at 1mL/kg/hr for 6 hours post-procedure
Arm/Group | 1, N-Acetylcysteine | 2, Sodium Bicarbonate
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/23
Other Adverse Events (participants affected / at risk) | 0/18 | 0/23

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed; Technical problems with measurement leading to unreliable or uninterpretable data. Rate of 72 hour Creatinine determination was poor.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No